CLINICAL TRIAL: NCT05210595
Title: The Early De-escalation Strategy With Ticagrelor 60 mg or 45 mg on Platelet Reactivity and Clinical Outcomes in Korean Patients With Acute Myocardial Infarction
Brief Title: Optimal Dosage of Ticagrelor in Korean Patients With AMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, Professor, Dept. of Cardiology Dong-A University Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOPE-TAILOR 2
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Acute Myocardial Infarction; Ticagrelor
Keywords: Ticagrelor; De-escalation Strategy; Korean
MeSH Terms: interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Clopidogrel 75 mg/day as maintenance dose
  Interventions: Drug: Clopidogrel 75 mg
- Treatment group 1 (Experimental): De-escalation strategy dose receive ticagrelor 60 mg twice daily
  Interventions: Drug: Ticagrelor 60mg
- Treatment group 2 (Experimental): De-escalation strategy dose receive ticagrelor 45 mg twice daily
  Interventions: Drug: Ticagrelor 45 mg

INTERVENTIONS:
Drug: Clopidogrel 75 mg — 75 mg/day as maintenance dose.
  Other Names: Plavix 75 mg
  Arms: Control group
Drug: Ticagrelor 60mg — In-hospital treatment with standard strategy ticagrelor 90mg twice daily, following de-escalation strategy ticagrelor 60 twice daily after discharge or post PCI 1 week.
  Other Names: Brilinta 60 mg
  Arms: Treatment group 1
Drug: Ticagrelor 45 mg — In-hospital treatment with standard strategy ticagrelor 90mg twice daily, following de-escalation strategy ticagrelor 45 twice daily after discharge or post PCI 1 week .
  Other Names: Brilinta 45 mg
  Arms: Treatment group 2

SUMMARY:
East Asian patients will be required optimal dose of newer P2Y12 inhibitor (ticagrelor) to determine the safer treatment and better outcome. Whether low dose of ticagrelorI is more adequate for clinical practice in Korea is unclear. Therefore, the investigators aim to evaluate efficacy and safety of low dose of ticagrelor in Acute Myocardial Infarction (AMI) undergoing percutaneous coronary intervention(PCI).

DETAILED DESCRIPTION:
In recent years, newer oral P2Y12 receptor blocker (ticagrelor) has been strong recommendations for management of patients with AMI undergoing (PCI). This drug provided more profound inhibitory effects than clopidogrel, which could lead to marked reduction in ischemic events, with relatively increase in bleeding complication, specific to low body weight, especially in women and East Asian patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients present with acute myocardial infarction undergoing PCI.
* Patients receiving ticagrelor; Male or female gender; Age 20-75 years.
* Patients provide written informed consent prior to enrollment.

Exclusion Criteria:

* Low body weight (<60kg).
* History of hemorrhagic stroke.
* History of upper gastrointestinal bleeding in recent 6 months.
* Bleeding tendency.
* Thrombocytopenia defined by platelet < 100,000/ml.
* Anemia defined by hemoglobin < 10 g/dl.
* Renal dysfunction defined as serum creatinine > 2.5 mg/dl.
* Severe hepatic dysfunction defined as serum transaminase > 3 times normal limit.
* Known severe chronic obstructive pulmonary disease or bradycardia (sick sinus syndrome (SSS) or high degree AV block without pacemaker protection).
* Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromycin.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimal platelet reactivity (OPR) rate | At 1 month
  OPR, indicate 85 to 208 for P2Y12 reaction units (PRU)

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | At 9 months
  MACCE: composite of cardiac death, non-fatal myocardial infarction, target lesion / vessel revascularization and stroke
Bleeding events | At 9 months.
  BARC: Bleeding Academic Research Consortium (BARC ≥2).

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, MD, Principal Investigator — Dong-A University Hospital
Locations (1):
- DongA University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No